CLINICAL TRIAL: NCT04036227
Title: A Phase I, Placebo-controlled, Double-blind, First-in-human Study to Investigate Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of GS-248 Solution in Healthy Subjects and Patients With Systemic Sclerosis (SSc)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GS-248
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gesynta Pharma AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-1001
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part I (SAD) Within each cohort, subjects will be randomised in a 3:1 ratio to receive either GS 248 (n=6) or placebo (n=2) in a blinded fashion.
  Part II (MAD) Within each cohort, subjects will be randomised in a 3:1 ratio to receive GS-248 (n=6) or placebo (n=2) in a blinded fashion.
Who Masked: Participant, Investigator
Masking Description: The study will be conducted in double-blind fashion and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
  GS-248 and the placebo are identical in appearance, taste and smell.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS-248 (Experimental): Part I (SAD): Single doses of 1 mg, 5 mg, 25 mg, 75 mg, 225 mg and 450 mg (planned doses)
  Part II (MAD): Multiple ascending doses for 10 days in four cohorts with planned doses of 25 mg, 75 mg, 225 mg and 450 mg. The doses will be finally selected based on results from Part I.
  Interventions: Drug: GS-248
- Placebo (Placebo Comparator): Matching placebo oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-248 — GS-248 oral solution
  Arms: GS-248
Drug: Placebo — Placebo oral solution with the same composition to match active drug
  Arms: Placebo

SUMMARY:
This is a First in Human (FIH), double-blinded, parallel-group, randomised, placebo-controlled study designed to evaluate the safety, tolerability, PK and PD of single and multiple ascending oral doses of GS-248 in healthy subjects.

DETAILED DESCRIPTION:
Part I (SAD); In the SAD part of the study, single oral doses of GS-248 will be administered in 6 sequential cohorts, each consisting of 8 subjects randomised to receive either GS 248 or placebo in a 3:1 ratio. The first 2 subjects in each cohort will be dosed in a sentinel fashion; 1 subject will receive GS-248 and the other will receive placebo as randomised. The subjects will be carefully monitored by clinical staff during and after dosing. Vital signs, safety laboratory and ECG will be checked at regular intervals.

Part II (MAD); The MAD part of the study will explore multiple ascending dosing of GS-248 administered for 10 days. The proposed starting dose is 25 mg/day. However, the starting dose as well as subsequent dose levels may be adjusted based on safety and PK evaluation in previous cohorts. GS-248 will be administered in 4 sequential cohorts, each of 8 subjects randomised to receive either GS 248 or placebo in a 3:1 ratio. The subjects will be carefully monitored by clinical staff during and after dosing. Vital signs, safety laboratory and ECG will be checked at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Male and female healthy subjects aged 18-70 years inclusive (Part I [SAD]) and 40-75 years inclusive (Part II [MAD])
3. Women of child bearing potential must practice abstinence or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy from at least 4 weeks prior to dose to 4 weeks after last dose. Their male partner must agree to use a condom during the same time frame. Women of non-childbearing potential are defined as pre-menopausal females who are sterilised or post-menopausal defined as 12 months of amenorrhea.

   Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence. Their female partner of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above).
4. Body mass index (BMI) ≥ 19 and ≤ 30 kg/m2.
5. Subjects must be in good health as determined by medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory assessments at the time of screening, as judged by the Investigator.

Exclusion Criteria:

1. Known allergy to any components of the GS-248 formulation.
2. Females who are breast feeding or plan to be pregnant.
3. Positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening and within 24 h prior to the first administration of Investigational Medicinal Product (IMP).
4. Use of corticosteroids (inhaled and systemic), NSAIDs (including e.g. coxibs and aspirin), antacids, Proton pump inhibitors (PPIs) or any medication that changes gastric pH within 2 weeks prior to the (first) administration of IMP.
5. Regular use of any prescribed or non-prescribed medication including analgesics, herbal remedies, vitamins and minerals within 2 weeks prior to the (first) administration of IMP, except hormonal contraception and occasional intake of paracetamol (maximum 2000 mg/day; and not exceeding 3000 mg/week) and nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
6. Inherited or acquired disorders of platelet function, bleeding or coagulation.
7. Presence of any clinically relevant acute or chronic disease that could interfere with the subject's safety during the clinical study or expose the subject to undue risk.
8. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

   * Systolic blood pressure <90 or >140 mmHg, or
   * Diastolic blood pressure <50 or >90 mmHg, or
   * Pulse <40 or >90 bpm
9. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV) 1 and/or 2 antibodies at screening.
10. Presence or history of drug and/or alcohol abuse and/or excessive intake of alcohol and/or history, or current use, of anabolic steroids, as judged by the Investigator.
11. Any positive result for drug abuse and/or alcohol at screening or on admission to the unit prior to administration of the IMP.
12. Participation in another clinical study with an experimental drug within 3 months before the administration of IMP.
13. Consumption of grapefruit or grapefruit juice within 14 days of study drug administration.
14. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
15. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma or resected benign colonic polyps.
16. Any planned major surgery within the duration of the study.
17. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
18. Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than 3 times per week is allowed before screening visit.
19. Regular excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages.
20. Intake of xanthine and/or taurine containing energy drinks within 2 days prior to screening.
21. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
22. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Folke Sjöberg, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from CTC's database of healthy volunteers and from advertising in media (including social media). Screening visits were performed at CTC research clinic.
  Part I (SAD): Recruitment period started 19JUN2019 and lasted until 15OCT2019. Part II (MAD): Recruitment period started in August 2019 (when first SAD cohorts had been completed) and lasted until 25NOV2019.
Pre-assignment Details: Part I (SAD): 92 subjects screened, 48 randomised to 6 dosing groups each of which included placebo. Did not meet the eligibility criteria=12, withdrew consent prior to randomisation=20, reserves=6, other reasons=6.
  Part II (MAD): 49 subjects screened, 24 randomised to 3 dosing groups each of which included placebo. Did not meet the eligibility criteria=11, withdrew consent prior to randomisation=9, reserve=1, other reasons=4.
Groups:
- Part I (SAD): 1 mg: Single dose (actual dose) of 1 mg GS-248 oral solution.
- Part I (SAD): 5 mg: Single dose (actual dose) of 5 mg GS-248 oral solution.
- Part I (SAD): 8 mg: Single dose (actual dose) of 8 mg GS-248 oral solution.
- Part I (SAD): 40 mg: Single dose (actual dose) of 40 mg GS-248 oral solution.
- Part I (SAD): 100 mg: Single dose (actual dose) of 100 mg GS-248 oral solution.
- Part I (SAD): 300 mg: Single dose (actual dose) of 300 mg GS-248 oral solution.
- Part I (SAD): Placebo; Part II (MAD): Placebo: Matching placebo oral solution
  Placebo: Placebo oral solution with the same composition to match active drug
- Part II (MAD): 20 mg: Multiple ascending doses for 10 days with actual dose of 20 mg. Dose were finally selected based on results from Part I.
- Part II (MAD): 60 mg: Multiple ascending doses for 10 days with actual dose of 60 mg.
- Part II (MAD): 180 mg: Multiple ascending doses for 10 days with actual dose of 180 mg.
Period: Part I (SAD): 1 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I (SAD): 5 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I (SAD): 8 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I (SAD): 40 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I (SAD): 100 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I (SAD): 300 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part I (SAD): Placebo
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II (MAD): 20 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II (MAD): 60 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II (MAD): 180 mg
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part II (MAD): Placebo
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I (SAD): 1 mg: Single dose of 1 mg GS-248 oral solution.
- Part I (SAD): 5 mg: Single dose of 5 mg GS-248 oral solution.
- Part I (SAD): 8 mg: Single dose of 8 mg GS-248 oral solution.
- Part I (SAD): 40 mg: Single dose of 40 mg GS-248 oral solution.
- Part I (SAD): 100 mg: Single dose of 100 mg GS-248 oral solution.
- Part I (SAD): 300 mg: Single dose of 300 mg GS-248 oral solution.
- Part I (SAD): Placebo: Single dose of matching placebo oral solution.
- Part II (MAD): 20 mg: Multiple ascending doses for 10 days with 20 mg.
- Part II (MAD): 60 mg: Multiple ascending doses for 10 days with 60 mg.
- Part II (MAD): 180 mg: Multiple ascending doses for 10 days with 180 mg.
- Part II (MAD): Placebo: Multiple ascending doses for 10 days with matching placebo oral solution.
- Total: Total of all reporting groups
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part I (SAD-cohorts) and Part II (MAD-cohorts) analysed separately.
  years
    Part I (SAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    Part I (SAD) | 40.7 (21.5) | 33.7 (9.8) | 36.8 (21.4) | 41.8 (15.9) | 50.7 (10.8) | 33.7 (13.0) | 32.4 (14.1) |  |  |  |  | 37.8 (15.8)
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD) |  |  |  |  |  |  |  | 56.7 (12.2) | 58.2 (11.0) | 58.2 (12.2) | 59.0 (13.9) | 58.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The demographics and baseline characteristics for subjects included in the different Part I (SAD) cohorts (dose level 1-300 mg) and Part II (MAD) cohorts (dose levels 20-180 mg) are presented separately since subjects were only included in one cohort.
  Participants
    Part I (SAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    Part I (SAD): Female | 2 | 3 | 1 | 3 | 4 | 4 | 3 |  |  |  |  | 20
    Part I (SAD): Male | 4 | 3 | 5 | 3 | 2 | 2 | 9 |  |  |  |  | 28
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD): Female |  |  |  |  |  |  |  | 4 | 4 | 4 | 3 | 15
    Part II (MAD): Male |  |  |  |  |  |  |  | 2 | 2 | 2 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The demographics and baseline characteristics for subjects included in the different Part I (SAD) cohorts (dose level 1-300 mg) and Part II (MAD) cohorts (dose levels 20-180 mg) are presented separately since subjects were only included in one cohort.
  Participants
    Part I (SAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    Part I (SAD): Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Part I (SAD): Not Hispanic or Latino | 6 | 6 | 6 | 5 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 47
    Part I (SAD): Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD): Hispanic or Latino |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part II (MAD): Not Hispanic or Latino |  |  |  |  |  |  |  | 6 | 6 | 6 | 6 | 24
    Part II (MAD): Unknown or Not Reported |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The demographics and baseline characteristics for subjects included in the different Part I (SAD) cohorts (dose level 1-300 mg) and Part II (MAD) cohorts (dose levels 20-180 mg) are presented separately since subjects were only included in one cohort.
  Participants
    part I (MAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    part I (MAD): American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    part I (MAD): Asian | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
    part I (MAD): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    part I (MAD): Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    part I (MAD): White | 4 | 5 | 6 | 6 | 6 | 6 | 11 | 0 | 0 | 0 | 0 | 44
    part I (MAD): More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    part I (MAD): Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD): American Indian or Alaska Native |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part II (MAD): Asian |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part II (MAD): Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part II (MAD): Black or African American |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part II (MAD): White |  |  |  |  |  |  |  | 6 | 6 | 6 | 6 | 24
    Part II (MAD): More than one race |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
    Part II (MAD): Unknown or Not Reported |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 72
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: The demographics and baseline characteristics for subjects included in the different Part I (SAD) cohorts (dose level 1-300 mg) and Part II (MAD) cohorts (dose levels 20-180 mg) are presented separately since subjects were only included in one cohort.
  kg/m^2
    Part I (SAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    Part I (SAD) | 22.3 (2.6) | 25.2 (3.9) | 25.2 (3.4) | 25.7 (3.4) | 26.0 (2.2) | 22.0 (2.0) | 24.0 (3.0) |  |  |  |  | 24.4 (3.2)
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD) |  |  |  |  |  |  |  | 26.0 (1.3) | 23.5 (2.7) | 24.3 (1.6) | 25.8 (3.5) | 24.9 (2.5)
Height [Mean (Standard Deviation); unit: cm] — Population: The demographics and baseline characteristics for subjects included in the different Part I (SAD) cohorts (dose level 1-300 mg) and Part II (MAD) cohorts (dose levels 20-180 mg) are presented separately since subjects were only included in one cohort.
  cm
    Part I (SAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    Part I (SAD) | 171.3 (13.6) | 169.0 (11.0) | 178.0 (4.4) | 176.7 (13.9) | 176.2 (9.6) | 173.3 (10.3) | 175.7 (10.4) |  |  |  |  | 174.1 (10.6)
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD) |  |  |  |  |  |  |  | 171.0 (11.9) | 171.7 (8.0) | 172.2 (6.8) | 176.0 (12.7) | 172.7 (9.7)
Weight [Mean (Standard Deviation); unit: kg] — Population: The demographics and baseline characteristics for subjects included in the different Part I (SAD) cohorts (dose level 1-300 mg) and Part II (MAD) cohorts (dose levels 20-180 mg) are presented separately since subjects were only included in one cohort.
  kg
    Part I (SAD): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 48
    Part I (SAD) | 65.7 (13.4) | 72.5 (16.9) | 79.8 (13.3) | 81.0 (18.0) | 81.0 (11.0) | 66.3 (8.2) | 74.7 (13.8) |  |  |  |  | 74.4 (14.5)
    Part II (MAD): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    Part II (MAD) |  |  |  |  |  |  |  | 76.2 (9.0) | 69.8 (11.9) | 72.3 (5.5) | 81.0 (17.2) | 74.8 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Events
Description: AEs were assessed as 'unlikely', 'possibly' or 'probably' related to the IMP. 'Possibly' and 'probably' were categorized as treatment related.
Time Frame: AEs were collected from the start of IMP administration until the end-of-study visit of each part, an average of 10 days in Part 1 (SAD) and 20 days in Part 2 (MAD).
Population: All subjects who have been randomised and received at least one dose of IMP.
Measure: Number; unit: Number of events
Groups:
- GS-248 1 mg (SAD): Part I; GS-248 1 mg SAD
- GS-248 5 mg (SAD): Part I; GS-248 5 mg SAD
- GS-248 8 mg (SAD): Part I; GS-248 8 mg SAD
- GS-248 40 mg (SAD): Part I; GS-248 40 mg SAD
- GS-248 100 mg (SAD): Part I; GS-248 100 mg SAD
- GS-248 300 mg (SAD): Part I; GS-248 300 mg SAD
- Placebo (SAD): Part I; Placebo (SAD)
- GS-248 20 mg (MAD): Part II; GS-248 20 mg MAD
- GS-248 60 mg (MAD): Part II; GS-248 60 mg MAD
- GS-248 180 mg (MAD): Part II; GS-248 180 mg MAD
- Placebo (MAD): Part II; Placebo (MAD)
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | Placebo (SAD) | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD) | Placebo (MAD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Number of events | 3 | 4 | 0 | 3 | 2 | 1 | 4 | 1 | 12 | 9 | 0

2. Primary Outcome: Clinically Significant Changes in ECG
Description: Single 12-lead ECG was recorded in supine position after 10 minutes of rest using an ECG machine. Heart rate and PQ/PR, QRS, QT and QTcF intervals were recorded. Ambulatory ECG telemetry was used for cardiac surveillance up to 24 h after IMP administration in the SAD part of the study.
Time Frame: 12-lead ECG was measured at pre-defined timepoints from the screening visit until the end-of-study visit, an average of 10 days in Part I (SAD) and 20 days in Part II (MAD).
Population: All subjects who have been randomised and received at least one dose of IMP.
Measure: Number; unit: Number of abnormal CS events
Groups:
- Placebo (SAD): Part I; Placebo SAD
- Placebo (MAD): Part II; Placebo MAD
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | Placebo (SAD) | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD) | Placebo (MAD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Number of abnormal CS events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Clinically Significant Changes in Vital Signs
Description: Systolic and diastolic blood pressure and pulse were measured in supine position after 10 minutes of rest. Body temperature was measured orally using a digital thermometer.
Time Frame: Vital signs was checked at pre-defined timepoints from the screening visit until the end-of-study visit, an average of 10 days in Part 1 (SAD) and 20 days in Part 2 (MAD).
Population: All subjects who have been randomised and received at least one dose of IMP.
Measure: Number; unit: Number of abnormal CS events
Groups:
- Total (SAD): All participants in Part I (SAD), both GS-248 and placebo.
- Total (MAD): All participants in Part II (MAD), both GS-248 and placebo.
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | Placebo (SAD) | Total (SAD) | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD) | Placebo (MAD) | Total (MAD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48 | 6 | 6 | 6 | 6 | 24
Number of abnormal CS events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Clinically Significant Changes in Safety Laboratory Parameters
Description: Blood samples for analysis of clinical chemistry, haematology and coagulation parameters.
Time Frame: Blood samples were collected at pre-defined timepoints from the screening visit until the end-of-study visit, an average of 10 days in Part I (SAD) and 20 days in Part II (MAD).
Population: All subjects who have been randomised and received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- GS-248 40 mg (SAD): Part I, GS-248 40 mg (SAD)
- GS-248 20 mg (MAD): Part II; GS-248 20 mg (MAD)
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | Placebo (SAD) | Total (SAD) | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD) | Placebo (MAD) | Total (MAD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48 | 6 | 6 | 6 | 6 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3

5. Primary Outcome: Clinically Significant Changes in Physical Examination
Description: A complete physical examination included assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities.
Time Frame: Physical examination was performed at pre-defined timepoints from the screening visit until the end-of- study visit, an average of 10 days in Part I (SAD) and 20 days in Part II (MAD).
Population: All subjects who have been randomised and received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- GS-248 5 mg (SAD): Part I; GS-248 5 mg (SAD)
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | Placebo (SAD) | Total (SAD) | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD) | Placebo (MAD) | Total (MAD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48 | 6 | 6 | 6 | 6 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2

6. Secondary Outcome: Cmax:
Description: Maximum plasma concentration.
Time Frame: SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose; MAD Day 1-3 (first dose) and Day 10-12 (last dose): pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose.
Population: All subjects who received at least one dose of the study drug and provided at least one evaluable plasma concentration profile without any AEs or protocol deviations judged to affect the PK analysis.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- GS-248 20 mg (MAD First Dose): Part II; GS-248 20 mg MAD Day 1-3 (first dose)
- GS-248 60 mg (MAD First Dose): Part II; GS-248 60 mg MAD Day 1-3 (first dose)
- GS-248 180 mg MAD (First Dose): Part II; GS-248 180 mg MAD Day 1-3 (first dose)
- GS-248 20 mg (MAD Last Dose): Part II; GS-248 20 mg MAD Day 10-12 (last dose)
- GS-248 60 mg (MAD Last Dose): Part II; GS-248 60 mg MAD Day 10-12 (last dose)
- GS-248 180 mg MAD (Last Dose): Part II; GS-248 180 mg MAD Day 10-12 (last dose)
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | GS-248 20 mg (MAD First Dose) | GS-248 60 mg (MAD First Dose) | GS-248 180 mg MAD (First Dose) | GS-248 20 mg (MAD Last Dose) | GS-248 60 mg (MAD Last Dose) | GS-248 180 mg MAD (Last Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
nmol/L | 1.247 (0.9537) | 8.975 (4.971) | 11.82 (4.365) | 145.3 (69.75) | 263.3 (65.07) | 818.3 (783.3) | 41.47 (18.45) | 231.8 (187.3) | 478.5 (310.0) | 43.93 (30.10) | 176.5 (83.04) | 903.0 (590.6)

7. Secondary Outcome: Tmax:
Description: Time to Cmax.
Time Frame: SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose; MAD: Day 1-3 (first dose) Day 10-12 (last dose): pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose.
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Groups:
- GS-248 180 mg (MAD First Dose): Part II; GS-248 180 mg MAD Day 1-3 (first dose)
- GS-248 180 mg (MAD Last Dose): Part II; GS-248 180 mg MAD Day 10-12 (last dose)
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | GS-248 20 mg (MAD First Dose) | GS-248 60 mg (MAD First Dose) | GS-248 180 mg (MAD First Dose) | GS-248 20 mg (MAD Last Dose) | GS-248 60 mg (MAD Last Dose) | GS-248 180 mg (MAD Last Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
hours | 1.500 [1.00 to 1.50] | 2.500 [1.50 to 3.00] | 1.000 [1.00 to 2.00] | 1.000 [0.500 to 1.50] | 1.000 [0.500 to 1.50] | 1.500 [1.00 to 2.00] | 1.000 [0.500 to 2.00] | 1.000 [0.500 to 1.00] | 1.108 [0.517 to 2.00] | 2.000 [1.00 to 2.00] | 1.000 [0.500 to 2.02] | 2.000 [1.02 to 2.05]

8. Secondary Outcome: T½:
Description: Terminal elimination half-life
Time Frame: SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose); MAD: Day 1-3 and Day 10-12: pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | GS-248 20 mg (MAD First Dose) | GS-248 60 mg (MAD First Dose) | GS-248 180 mg (MAD First Dose) | GS-248 20 mg (MAD Last Dose) | GS-248 60 mg (MAD Last Dose) | GS-248 180 mg (MAD Last Dose)
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
hours | 4.539 (2.435) | 1.089 (0.1879) | 1.660 (0.3684) | 9.220 (6.697) | 9.513 (3.683) | 11.14 (1.630) | 3.469 (2.073) | 6.705 (3.120) | 11.86 (10.76) | 6.504 (3.980) | 18.00 (8.750) | 15.01 (5.225)

9. Secondary Outcome: AUC0-t:
Description: Area under the concentration time curve from the time of dosing to the time of the last observation.
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*nmol/L
Groups:
- GS-248 1 mg (SAD): Part I; GS-248 1 mg (SAD).
- GS-248 8 mg (SAD): Part I, GS-248 8 mg (SAD)
- GS-248 40 mg (SAD): Part I; GS-248 40 mg (SAD)
- GS-248 100 mg (SAD): Part I; GS-248 100 mg (SAD).
- GS-248 300 mg (SAD): Part I; GS-248 300 mg (SAD)
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | GS-248 20 mg (MAD First Dose) | GS-248 60 mg (MAD First Dose) | GS-248 180 mg (MAD First Dose) | GS-248 20 mg (MAD Last Dose) | GS-248 60 mg (MAD Last Dose) | GS-248 180 mg (MAD Last Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
h*nmol/L | 2.437 (1.846) | 30.57 (22.88) | 39.08 (13.40) | 478.6 (285.3) | 879.8 (380.0) | 2667 (2850) | 180.1 (75.75) | 655.8 (473.7) | 1735 (1164) | 211.0 (115.5) | 650.5 (267.2) | 4798 (3702)

10. Secondary Outcome: AUC 0-inf
Description: Area under the curve from time 0 to infinity.
Time Frame: SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD)
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6
h*nmol/L | 8.542 (0.8438) | 40.22 (24.62) | 41.77 (13.80) | 489.3 (282.3) | 894.7 (380.8) | 2713 (2906)

11. Secondary Outcome: AUCss
Description: Area under the plasma concentration curve during a dosing interval at steady state.
Time Frame: MAD: Day 10-12: pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose.
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD)
Number analyzed (Participants) | 6 | 6 | 5
h*nmol/L | 205.9 (103.4) | 604.6 (233.1) | 4046 (2823)

12. Secondary Outcome: Clearance (CL)/F:
Description: Apparent total body clearance following extravascular administration.
Time Frame: SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose); MAD Day 1-3 and Day 10-12: pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- GS-248 20 mg (MAD First Dose): Part I; GS-248 20 mg MAD Day 1-3 (first dose).
- GS-248 60 mg (MAD First Dose): Part I; GS-248 60 mg MAD Day 1-3 (first dose).
- GS-248 180 mg (MAD First Dose): Part I; GS-248 180 mg MAD Day 1-3 (first dose).
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | GS-248 20 mg (MAD First Dose) | GS-248 60 mg (MAD First Dose) | GS-248 180 mg (MAD First Dose) | GS-248 20 mg (MAD Last Dose) | GS-248 60 mg (MAD Last Dose) | GS-248 180 mg (MAD Last Dose)
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
L/h | 173.7 (17.51) | 228.2 (102.7) | 304.8 (83.80) | 161.4 (92.39) | 184.8 (58.74) | 318.2 (223.4) | 187.0 (79.05) | 190.2 (109.1) | 181.2 (101.4) | 175.4 (81.81) | 166.2 (63.62) | 97.59 (74.02)

13. Secondary Outcome: Vz/F:
Description: Apparent volume of distribution following extravascular administration
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | GS-248 1 mg (SAD) | GS-248 5 mg (SAD) | GS-248 8 mg (SAD) | GS-248 40 mg (SAD) | GS-248 100 mg (SAD) | GS-248 300 mg (SAD) | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD)
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 5
L | 1097 (516.4) | 341.9 (120.5) | 719.7 (192.1) | 2117 (2445) | 2378 (918.8) | 4856 (3394) | 1354 (392.3) | 3945 (1685) | 2157 (2139)

14. Secondary Outcome: Accumulation Ratio AUC 0-ss
Time Frame: MAD: Day 1-3 and Day 10-12: pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GS-248 20 mg (MAD) | GS-248 60 mg (MAD) | GS-248 180 mg (MAD)
Number analyzed (Participants) | 6 | 6 | 5
ratio | 1.148 (0.3148) | 1.171 (0.5541) | 2.390 (1.135)

15. Other Pre Specified Outcome: mPGES-1 Activity
Description: Ex vivo determination of mPGES-1 activity in a Whole Blood Assay (WBA) measured as percent change from baseline of Prostaglandin E2 (PGE2) levels after lipopolysaccharide (LPS) stimulation.
Time Frame: At 24h after first dose Day 1 and at 24 hours after last dose Day 10.
Population: All subjects who were randomised, received at least one dose of IMP and who had at least one post-baseline assessment of efficacy data.
Measure: Mean (Standard Deviation); unit: Relative change from baseline (%)
Groups:
- Day 1 (SAD): 5 mg: 24 hours after dose Day 1 (SAD): Single dose of 5 mg GS-248.
- Day 1 (SAD): 40 mg: 24 hours after dose Day 1 (SAD): 40 mg GS-248.
- Day 1 (SAD): 100 mg: 24 hours after dose Day 1 (SAD): 100 mg GS-248.
- Day 1 (SAD): 300 mg: 24 hours after dose Day 1 (SAD): 300 mg GS-248.
- Day 1 (MAD): 20 mg: 24 hours after dose Day 1 (MAD): 20 mg GS-248.
- Day 1 (MAD): 60 mg: 24 hours after dose Day 1 (MAD): 60 mg GS-248.
- Day 1 (MAD): 180 mg: 24 hours after dose Day 1 (MAD): 180 mg GS-248.
- Day 1 (SAD and MAD): Placebo: 24 hours after dose Day 1 (SAD and MAD): Placebo.
- Day 10 (MAD): 20 mg: 24 hours after last dose, administered Day 10, (MAD): 20 mg GS-248.
- Day 10 (MAD): 60 mg: 24 hours after last dose administered Day 10 (MAD): 60 mg GS-248.
- Day 10 (MAD): 180 mg: 24 hours after last dose administered Day 10 (MAD): 180 mg GS-248.
- Day 10 (MAD): Placebo: 24 hours after last dose administered Day 10 (MAD): Placebo
Arm/Group | Day 1 (SAD): 5 mg | Day 1 (SAD): 40 mg | Day 1 (SAD): 100 mg | Day 1 (SAD): 300 mg | Day 1 (MAD): 20 mg | Day 1 (MAD): 60 mg | Day 1 (MAD): 180 mg | Day 1 (SAD and MAD): Placebo | Day 10 (MAD): 20 mg | Day 10 (MAD): 60 mg | Day 10 (MAD): 180 mg | Day 10 (MAD): Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 5 | 6
Relative change from baseline (%) | 7.2 (98.8) | -97.1 (12.1) | -108.3 (11.5) | -105.2 (11.6) | -65.9 (20.2) | -94.9 (9.3) | -104.3 (6.8) | 9.8 (59.6) | -86.9 (26.8) | -104.3 (13.9) | -109.8 (7.8) | 18.6 (57.7)

ADVERSE EVENTS:
Time Frame: AEs (including serious AEs [SAEs]) were collected from the start of IMP application until the end-of- study visit of each part, an average of 10 days in Part I (SAD) and 20 days in Part II (MAD).
Description: The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. AEs were assessed as unlikely, possibly or probably related to the IMP
Groups:
- Part II (MAD): 20 mg: Multiple ascending doses for 10 days with actual dose of 20 mg.
Arm/Group | Part I (SAD): 1 mg | Part I (SAD): 5 mg | Part I (SAD): 8 mg | Part I (SAD): 40 mg | Part I (SAD): 100 mg | Part I (SAD): 300 mg | Part I (SAD): Placebo | Part II (MAD): 20 mg | Part II (MAD): 60 mg | Part II (MAD): 180 mg | Part II (MAD): Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 0/6 | 1/6 | 3/6 | 4/6 | 5/12 | 5/6 | 5/6 | 5/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I (SAD): 1 mg (N=6) | Part I (SAD): 5 mg (N=6) | Part I (SAD): 8 mg (N=6) | Part I (SAD): 40 mg (N=6) | Part I (SAD): 100 mg (N=6) | Part I (SAD): 300 mg (N=6) | Part I (SAD): Placebo (N=12) | Part II (MAD): 20 mg (N=6) | Part II (MAD): 60 mg (N=6) | Part II (MAD): 180 mg (N=6) | Part II (MAD): Placebo (N=6)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 1 (1) | 2 (3) | 1 (1) | 1 (1) — Headache
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Abdominal pain
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Constipation
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Lip dry
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Nausea
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Paraesthesia oral
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Vomiting
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dyspnoea
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Nasopharyngitis
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Oropharyngeal pain
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Malaise
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Pyrexia
Vessel puncture site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Vessel puncture site thrombosis
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Influenza
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Nasopharyngitis
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Decreased appetite
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dysuria
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dysmenorrhoea
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hyperhidrosis
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hot flush
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Abdominal distension
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) — Diarrhoea
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) — Flatulence
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Toothache
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Dermatitis contact
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hyperhidrosis
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pruritus
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Rash
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Rash maculo-papular
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Swelling face
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Oropharyngeal pain
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Fatigue
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Peripheral swelling
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Rhinitis
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Anaemia
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Atrial fibrillation
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Muscular weakness
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Myalgia
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Ear discomfort
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Tinnitus
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Eye pruritus
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Aspartate aminotransferase increased
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Glucose tolerance impaired

LIMITATIONS AND CAVEATS:
Part I=SAD was completed in full. Part II=MAD was completed after three of four cohorts. Reason: Systemic exposure of GS-248 was considered sufficiently high after 3 MAD cohorts.

Part III= Systemic sclerosis patients was cancelled. Reason: Decision by Sponsor that performing this part would not add scientific value to the development programme for GS-248.

Part IV=Celecoxib was completed in full. Only celecoxib given in this exploratory comparison and thus results excluded in result section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any confidential information relating to the IMP or the study, including any data and results from the study, will be the exclusive property of the Sponsor. The Investigator and any other persons involved in the study are responsible for protecting the confidentiality of this proprietary information belonging to the Sponsor. The results from this study may be submitted for publication at the discretion of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT04036227/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT04036227/SAP_001.pdf